CLINICAL TRIAL: NCT05173142
Title: A Phase Ib/II Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of HMPL-453 (FGFR Inhibitor) Combined With Chemotherapy or Anti-PD-1 Antibody in Patients With Advanced Solid Tumors
Brief Title: HMPL-453 (FGFR Inhibitor) in Combination With Chemotherapy or Anti-PD-1 Antibody in Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021-453-00CH1
Record Dates: First submitted 2021-10-31; First posted 2021-12-29 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Solid Tumor
Keywords: HMPL-453, FGFR, PD-1,IHCC, ICC, gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gemcitabine; Cisplatin; toripalimab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dose escalation phase of HMPL-453 monotherapy or combination therapy (Experimental): HMPL-453 monotherapy or combination therapy
  Interventions: Drug: HMPL-453; Drug: gemcitabine and cisplatin; Drug: toripalimab
- indication specific dose expansion phase of HMPL-453 combination therapy (Experimental): HMPL-453 combined with chemotherapy or anti-PD-1 antibody, in patients with IHCC, G/GEJ, or UC harboring specific FGFR gene alterations
  Interventions: Drug: HMPL-453; Drug: gemcitabine and cisplatin; Drug: toripalimab; Drug: Docetaxel

INTERVENTIONS:
Drug: HMPL-453 — HMPL-453 administered orally.
Drug: gemcitabine and cisplatin — Gemcitabine and Cisplatin administered intravenously.
Drug: toripalimab — Toripalimab administered intravenously.
Drug: Docetaxel — Docetaxel administered intravenously.
  Arms: indication specific dose expansion phase of HMPL-453 combination therapy

SUMMARY:
This is a phase Ib/II clinical study designed to evaluate the safety, tolerability, and preliminary efficacy of HMPL-453 combined with chemotherapy or anti-PD-1 antibody in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The study includes a dose escalation phase and a dose-expansion phase.

Patients with advanced solid tumor will be enrolled in the dose escalation phase to assess the tolerability, safety, and PK profile of HMPL-453 monotherapy or combination therapy.

Patients with specific types of advanced or metastatic tumors harboring certain FGFR gene alterations will be enrolled in the dose expansion phase to assess the preliminary efficacy of HMPL-453 combination therapy.

ELIGIBILITY:
Inclusion Criteria

* Dose escalation phase: patients with histologically or cytologically confirmed locally advanced or metastatic solid tumor who progressed on or are intolerant of standard therapy;
* Dose expansion phase: patients with UC, GC/GEJ, or IHCC harboring specific FGFR gene alterations;
* Age 18 to 75 years;
* Those who are able to give written informed consent, and able to comply with protocol-specified visits and related procedures;
* Ability to swallow study drug;
* ECOG PS of 0 or 1;
* Measurable lesion according to RECIST v1.1, refer to the protocol;
* Adequate organ and bone marrow function;
* Life expectancy ≥ 12 weeks;
* Female patients or male patients with partners of childbearing potential must take effective contraceptive measures per the protocol.

Exclusion Criteria

* Patients who previously received selective FGFR targeting therapy;
* Concurrent participation in another interventional clinical study, excluding those in the follow-up period and have not recently received investigational intervention;
* Current or previous history of central nervous system (CNS) metastases；
* Current or previous history of retinal detachment；
* Known history of primary immunodeficiency;
* Female patients who are pregnant or lactating；
* Patients who in the opinion of the investigator may be unsuitable for participating in the study;
* Patients with acute or chronic active hepatitis B or C infection;
* Known human immunodeficiency virus (HIV) infection and syphilis infection；
* Clinically significant cardiovascular disease such as congestive heart failure or arrhythmia；
* Uncontrolled hypertension despite optimal medical management；
* Received live vaccine within 30 days before the first dose of study drug(s);
* Those who have undergone major surgical procedures (craniotomy, thoracotomy or laparotomy) within 4 weeks prior to the first study treatment or who are expected to be in need of major surgery; those with unhealed wounds, ulcers or fractures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2022-01-22 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability(Incidence and severity of adverse events (AEs)) | 6 months after the last patient enrolled
  DLT, TEAEs and SAEs
Preliminary efficacy/Objective response rate (ORR) | up to 2 years
  Objective response rate (ORR) in patients with the selected tumors along with certain FGFR gene alterations

SECONDARY OUTCOMES:
Efficacy/Progression-free survival (PFS) | up to 2 years
  the duration between the enrollment date and the first disease progression (PD) or death (whichever comes first).
disease control rate (DCR) | up to 2 years
  The incidence of complete response, partial response and stable disease
time to response (TTR) | up to 2 years
  The period from the date of enrollment to the date when the criteria for complete response or partial response was first measured (first record shall prevail).
duration of response (DoR） | up to 2 years
  The duration between the date the criteria for complete response or partial response was first measured (first record shall prevail) and the date of disease recurrence or progression as objectively recorded
overall survival (OS) | up to 2 years
  The period from date of enrollment to date of death

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China